CLINICAL TRIAL: NCT00207233
Title: Use of MCT Oil for Enhancement of Weight Loss and Glycemic Control in Obese Diabetic Patients 2002-292G
Brief Title: Use of MCT Oil for Enhancement of Weight Loss and Glycemic Control in Obese Diabetic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Caroline Apovian, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-22398
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2009-02

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
Keywords: Weight loss; MCT oil hypocaloric liquid diet; LCT oil hypocaloric liquid diet; Gastric Bypass
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Will receive MCT study oil to supplement into liquid meal replacements.
  Interventions: Behavioral: MCT oil hypocaloric liquid diet; Procedure: Subcutaneous abdominal adipose tissue biopsy
- 2 (Placebo Comparator): Will receive LCT oil to supplement into their liquid meal replacements.
  Interventions: Behavioral: LCT hypocaloric liquid diet; Procedure: Subcutaneous abdominal adipose tissue biopsy

INTERVENTIONS:
Behavioral: MCT oil hypocaloric liquid diet — The MCT diet will consist of 5 liquid meals using a commercial product (HMR 800 Health Management Resources, Inc.; 160 kcal/shake) plus 34 grams MCT oil (Life Enhancement Products, Inc. Petaluna, CA; 8.3 kcal/gm) added per day to the HMR shakes.
  The intervention will last 3 months. After the first 6 weeks you will be assessed for 5% weight loss. If reach this weight change you will continue on the same intervention for another 6 weeks. Those who do not lose 5% of their baseline weight will be withdrawn from the study.
  Arms: 1
Behavioral: LCT hypocaloric liquid diet — The LCT diet will consist of 5 liquid meals using a commercial product (HMR 800 Health Management Resources, Inc.; 160 kcal/shake) plus 31.5 grams LCT oil (corn oil; 9 kcal/gm) per day. Both diets will be isocaloric (1083 kcal/day) consisting of 38% CHO, 28% pro, 34% fat.
  The intervention will last 3 months. After the first 6 weeks you will be assessed for 5% weight loss. If reach this weight change you will continue on the same intervention for another 6 weeks. Those who do not lose 5% of their baseline weight will be withdrawn from the study.
  Arms: 2
Procedure: Subcutaneous abdominal adipose tissue biopsy — Subcutaneous adipose tissue biopsies from human subjects will provide tissue samples for ex vivo analysis of adipocytokine production and cell size. Subcutaneous adipose tissue will be sampled by needle biopsy at the suprailiac crest skinfold using standard sterile technique. After a 10 cm area is isolated, cleaned and anesthetized with 1% lidocaine, a small cutaneous incision (1 cm) will be performed. A 50 cc syringe with a 19-gauge needle will be used to aspirate approximately 150 mg of adipose tissue which will require 2 to 6 passes of the needle. Sutures will be used to close the skin incision and a dry sterile dressing applied.
  This will be performed at baseline, 6 weeks, and 12 weeks.

SUMMARY:
Phase I, 6 weeks: Intensive weight loss 42 obese subjects with type 2 diabetes mellitus or impaired fasting glucose (FBS greater than 100 mg/dl) and a patient at the Nutrition and Weight Management Center at Boston Medical Center will be randomized to receive either an MCT-based or LCT-based liquid diet for a 6 week period (Phase I) to establish compliance followed by a second 6 week period (Phase II). These diets will be isocaloric (1083 kcal/day) and identical except for the quality of the fat. The intervention will be double blinded. The MCT diet will consist of 5 liquid meals using a commercial product plus 34 grams MCT oil (Life Enhancement Products, Inc. Petaluna, CA; 8.3 kcal/gm) added per day to the HMR shakes. The LCT diet will utilize 5 HMR shakes plus 31.5 grams LCT oil (corn oil; 9 kcal/gm) per day. Patients in both groups will be given a list of supplemental foods that are suitable for the study. They may choose to eat up to an additional 400 kcal per day from this list and will be asked to add these to their food records for monitoring of their caloric intake. A dietitian will instruct subjects at a baseline visit on behavior modification and a moderate physical activity program. Baseline testing includes the following: Body composition by DEXA (Hologic); Subcutaneous abdominal adipose tissue biopsy; blood work. Subjects who do not lose 5% of their baseline weight by the end of Phase I will be withdrawn from the study. If subjects do not lose 5% in Phase I, they will be considered inappropriate for a liquid diet, and therefore for the study, and will be discontinued from the study.

Phase II, 6 weeks: Continued weight loss program during phase II, subjects will be maintained on the same diet, supplements and exercise program. Once patients enter Phase II, all baseline lab measurements will be repeated. Needle biopsies of subcutaneous abdominal adipose tissue will be obtained at the beginning and at at the end of Phase II. Finger-stick blood glucose levels will be checked weekly. At the end of Phase II, and of the study, fasting blood work will be obtained. At the end of Phase II, the following procedures will be performed: Subcutaneous abdominal adipose tissue biopsy (total = 3). Body composition by DEXA (Hologic) (total = 2).

DETAILED DESCRIPTION:
Phase I, 6 weeks: Intensive weight loss forty-two obese subjects with type 2 diabetes mellitus or impaired fasting glucose (FBS greater than 100 mg/dl) will be randomized to receive either an MCT-based or LCT-based liquid diet for a 6 week period (Phase I) to establish compliance followed by a second 6 week period (Phase II). These diets will be isocaloric (1083 kcal/day) and identical except for the quality of the fat . The intervention will be double blinded. The MCT diet will consist of 5 liquid meals using a commercial product (HMR 800 Health Management Resources, Inc.; 160 kcal/shake) plus 34 grams MCT oil (Life Enhancement Products, Inc. Petaluna, CA; 8.3 kcal/gm) added per day to the HMR shakes. The LCT diet will utilize 5 HMR shakes plus 31.5 grams LCT oil (corn oil; 9 kcal/gm) per day. Patients in both groups will be given a list of supplemental foods that are suitable for the study. They may choose to eat up to an additional 400 kcal per day from this list and will be asked to add these to their food records for monitoring of their caloric intake. A dietitian will instruct subjects at a baseline visit on behavior modification and a moderate physical activity program of walking for 30 minutes five times per week. Participants will complete food and exercise logs that will be analyzed by the study staff. Baseline testing includes the following: Body composition by DEXA (Hologic); Subcutaneous abdominal adipose tissue biopsy; blood for CBC, basic metabolic panel, LFT, TSH, C-reactive protein, HOMA-IR, fasting glucose, insulin, lipids (total cholesterol, HDL, LDL, triacyglycerol), hemoglobin A1c, hydroxybutyrate, free fatty acids, leptin, adiponectin, TNF-alpha, and PAI-1. For measuring dietary compliance throughout the entire study, three consecutive daily dietary records (two week day and one weekend day) will be analyzed each week by a registered dietitian using the Minnesota Nutrient Database. Subjects who do not lose 5% body weight by the end of Phase I will be withdrawn from the study. If subjects do not lose 5% in Phase I, they will be considered inappropriate for a liquid diet, and therefore for the study, and will be discontinued from the study.

Phase II, 6 weeks: Continued weight loss program During phase II, subjects will be maintained on the same diet, supplements and exercise program.Once patients enter Phase II, all baseline lab measurements will be repeated. Needle biopsies of subcutaneous abdominal adipose tissue will be obtained at the beginning and at at the end of Phase II. Finger-stick blood glucose levels will be checked weekly. At the end of Phase II, and of the study, the following data will be collected: Lab data: CBC, basic metabolic panel, LFT, TSH, C-reactive protein, fasting blood glucose, insulin, HOMA-IR, lipids (total cholesterol, HDL, LDL, triacyglycerol), HbA1c, hydroxybutyrate, FFA, leptin, adiponectin, TNF-alpha, and PAI-1 levels. At the end of Phase II, the following procedures will be performed: Subcutaneous abdominal adipose tissue biopsy (total = 3) ;. Body composition by DEXA (Hologic) (total = 2).

ELIGIBILITY:
Inclusion Criteria:

* Patient of the Nutrition and Weight Management Center at Boston Medical Center
* Obese ( BMI equal or greater to 30 kg/m2
* Men and women
* Age more than or equal to 18 years
* Type 2 diabetes mellitus controlled by diet or use of Metformin or Impaired fasting glucose (FBS more than or equal to 100 mg/dl)
* Only diet-controlled diabetics or those on Metformin will be considered since all classes of anti-diabetic agents have different effects on appetite and body weight, which may confound the interpretation of study results.

Exclusion Criteria:

* Currently not a patient at the Nutrition and Weight Management Center at Boston Medical Center
* Need for oral anti-diabetic agents (other than Metformin)
* Abnormal thyroid status: hyperthyroidism or hypothyroidism (TSH less than 0.5 or more than 5.0)
* Significant liver disease (bilirubin more than or equal to 2.0 or liver enzyme more than 3 times upper limited of normal range)
* Significant renal disease (creatinine more than or equal to 2.0)
* On the following medications known to affect carbohydrate and lipid metabolism: steroids, Beta adrenergic blockers, diuretics, insulin, and hypolipidemic agents
* Use of prescription or over the counter weight loss medications
* Weight loss of >5% or more in the last three (3) months
* Anorexia nervosa or bulimia nervosa
* Pregnancy or lactation
* Significant lactose intolerance
* Significant egg allergy
* History of drug or alcohol addiction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2004-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Weight change | 3 months
Waist circumference change | 3 months
Glycemic control | 3 months
Change in expression of selected adipocyte metabolic genes | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Apovian, MD, Principal Investigator — Boston University; James Kirkland, MD,PhD, Study Chair — Boston University; Peter Burke, MD, Study Chair — Boston University; Wen Guo, PhD, Study Chair — Boston University; Diana Cullum-Dugan, RD.LD, Study Chair — Boston University; Marie McDonnell, MD, Study Chair — Boston University; Donald Hess, MD, Study Chair — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Kuczmarski RJ, Flegal KM, Campbell SM, Johnson CL. Increasing prevalence of overweight among US adults. The National Health and Nutrition Examination Surveys, 1960 to 1991. JAMA. 1994 Jul 20;272(3):205-11. doi: 10.1001/jama.272.3.205. PMID 8022039
- [Background] Galuska DA, Serdula M, Pamuk E, Siegel PZ, Byers T. Trends in overweight among US adults from 1987 to 1993: a multistate telephone survey. Am J Public Health. 1996 Dec;86(12):1729-35. doi: 10.2105/ajph.86.12.1729. PMID 9003129
- [Background] Tuomilehto J, Wolf E. Primary prevention of diabetes mellitus. Diabetes Care. 1987 Mar-Apr;10(2):238-48. doi: 10.2337/diacare.10.2.238. PMID 3556107
- [Background] Wing RR. Use of very-low-calorie diets in the treatment of obese persons with non-insulin-dependent diabetes mellitus. J Am Diet Assoc. 1995 May;95(5):569-72; quiz 573-4. doi: 10.1016/S0002-8223(95)00155-7. PMID 7722192
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] St-Onge MP, Jones PJ. Physiological effects of medium-chain triglycerides: potential agents in the prevention of obesity. J Nutr. 2002 Mar;132(3):329-32. doi: 10.1093/jn/132.3.329. PMID 11880549
- [Background] Babayan VK. Medium chain triglycerides and structured lipids. Lipids. 1987 Jun;22(6):417-20. doi: 10.1007/BF02537271. PMID 3112486
- [Background] Lasekan JB, Rivera J, Hirvonen MD, Keesey RE, Ney DM. Energy expenditure in rats maintained with intravenous or intragastric infusion of total parenteral nutrition solutions containing medium- or long-chain triglyceride emulsions. J Nutr. 1992 Jul;122(7):1483-92. doi: 10.1093/jn/122.7.1483. PMID 1619475
- [Background] Bray GA, Lee M, Bray TL. Weight gain of rats fed medium-chain triglycerides is less than rats fed long-chain triglycerides. Int J Obes. 1980;4(1):27-32. PMID 7390698
- [Background] Geliebter A, Torbay N, Bracco EF, Hashim SA, Van Itallie TB. Overfeeding with medium-chain triglyceride diet results in diminished deposition of fat. Am J Clin Nutr. 1983 Jan;37(1):1-4. doi: 10.1093/ajcn/37.1.1. PMID 6849272
- [Background] Scalfi L, Coltorti A, Contaldo F. Postprandial thermogenesis in lean and obese subjects after meals supplemented with medium-chain and long-chain triglycerides. Am J Clin Nutr. 1991 May;53(5):1130-3. doi: 10.1093/ajcn/53.5.1130. PMID 2021124